CLINICAL TRIAL: NCT07394270
Title: Effect of Add-on L-Arginine Therapy on Clinical Outcome of Heart Failure Patients: A Randomized- Controlled Trial
Brief Title: Effect of Add-on L-Arginine Therapy on Heart Failure Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: German University in Cairo (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Araby, Msc., German University in Cairo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPH-2025-07-MHS
Record Dates: First submitted 2025-12-23; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure
Keywords: Heart failure; Drug repurposing; L-Arginine; Add-on therapy; HFrEF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-Arginine Arm (Active Comparator): Patients in this arm will be administered 6 gm L-arginine per day
  Interventions: Drug: L-Arginine Powder
- Placebo Arm (Placebo Comparator): Patients in this arm will take 6 gm placebo per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-Arginine Powder — L-arginine 3 gm sachets are used twice daily
  Arms: L-Arginine Arm
Drug: Placebo — 2 sachets of placebo are administered per day
  Arms: Placebo Arm

SUMMARY:
Heart failure is considered one of the greatest challenges globally. There are various treatment strategies for heart failure. L-Arginine is an amino acid that was found to have beneficial effect on vasculature. This study aims to study the benefits and side effects of using L-arginine on the patients with ejection fraction <40%

ELIGIBILITY:
Inclusion Criteria:

* Patients with EF <40%
* eGFR >30 mL/min/1.73 m2
* Stable patients
* Capable and willing to provide written consent

Exclusion Criteria:

* Patients with implantable cardioverter-defibrillator
* Pregnant or lactating fmeales
* Patients with a history of sensitivity to L-Arginine or any of the excipients
* Acute heart failure patients
* Patients use L-arginine supplementation.
* Patients with active herpes disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change of Global longitudinal strain value (GLS) of HF patients from the baseline | 6 weeks

SECONDARY OUTCOMES:
Change of heart failure symptoms as determined by NYHA classification from baseline | 6 weeks
Change of the functional abilities (ECG) of the patients as determined by the exercise test from baseline | 6 weeks
Changes in biomarkers of heart failure as determined by the difference in NT-proBNP levels from baseline | 6 weeks
Change in quality of life between 2 groups as determined by Minnesota Living with Heart Failure questionnaire | 6 weeks
Safety profile of the L-Arginine as determined by the change in the mean arterial pressure (MAP) between the 2 groups | 6 weeks
Change in biomarkers of endothelial dysfunction as determined by the difference in levels of endothelin-1 | 6 weeks
Change in biomarkers of endothelial dysfunction as determined by the difference in levels of Asymmetric dimethylarginine (ADMA) | 6 weeks
Safety profile of the L-Arginine as determined by the change in the heart rate (HR) between the 2 groups | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No